CLINICAL TRIAL: NCT04023201
Title: Nocturnal Symptoms and Quality of Life in Patients With Parkinson's Disease in Shanghai
Acronym: NQPDSH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XHEC-C-2019-094
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parkinson's disease patients: Parkinson's disease patients with or without nocturnal symptoms
  Interventions: Other: Nocturnal symptoms

INTERVENTIONS:
Other: Nocturnal symptoms — Parkinson's disease patients with or without nocturnal symptoms

SUMMARY:
This is a cross-sectional, retrospective clinical observation study focusing on the incidence and influencing factors of nocturnal symptoms in patients with Parkinson's disease.

DETAILED DESCRIPTION:
This study was a cross-sectional, retrospective clinical observation study investigating the incidence and influencing factors of nocturnal symptoms in patients with Parkinson's disease through the Parkinson's disease sleep-related scale. At the same time, the effects of nocturnal symptoms on the quality of life of patients with Parkinson's disease were studied. About 1,500 Parkinson's patients will be recruited into the study who come from Shanghai, China.

ELIGIBILITY:
Inclusion Criteria:

1. Parkinson's disease patients diagnosed according to the diagnostic criteria of MDS
2. Signing informed consent

Exclusion Criteria:

1. clinically suspected Parkinson's disease, has not been diagnosed;
2. suspected or diagnosed as secondary Parkinson's syndrome (vascular, drug, traumatic, encephalitis, toxic, etc.);
3. suspected or diagnosed as atypical Parkinson's syndrome (progressive supranuclear palsy, multiple system atrophy, cortical basal ganglia degeneration, etc.);
4. There is a clear history of stroke, moderate to severe traumatic brain injury, hydrocephalus, brain surgery or history of brain tumors;
5. severe cognitive impairment or psychiatric symptoms;
6. Can not cooperate with the completion of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Parkinson's disease patients diagnosed according to the diagnostic criteria of MDS
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2019-07-03 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
nocturnal symptoms in patients with Parkinson's disease | January 31, 2020
  the incidence and influencing factors of nocturnal symptoms in patients with Parkinson's disease

CONTACTS AND LOCATIONS:
Overall Officials: Zhenguo Liu, Doctor, Study Chair — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Grandas F, Iranzo A. Nocturnal problems occurring in Parkinson's disease. Neurology. 2004 Oct 26;63(8 Suppl 3):S8-11. doi: 10.1212/wnl.63.8_suppl_3.s8. PMID 15505143